CLINICAL TRIAL: NCT01230710
Title: A Multi-centre, Open-label, Phase IV, Interventional Study to Evaluate the Efficacy of Erlotinib (Tarceva®) Following 4 Cycles of Platinum-based Chemotherapy in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Who Have Not Experienced Disease Progression or Unacceptable Toxicity During Chemotherapy
Brief Title: A Study of Tarceva (Erlotinib) in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer Following 4 Cycles of Platinum-based Chemotherapy Without Disease Progression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25478
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Erlotinib (Experimental): Participants received erlotinib 150 mg orally once a day for 48 weeks.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib was supplied as tablets.
  Other Names: Tarceva

SUMMARY:
This open-label, single-arm study will evaluate the safety and efficacy of Tarceva (erlotinib) in patients with locally advanced or metastatic non-small cell lung cancer who have completed 4 cycles of standard platinum-based chemotherapy without progression. Patients will receive Tarceva at a dose of 150 mg orally daily until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Histologically documented non-small cell lung cancer (NSCLC).
* Locally advanced or recurrent (Stage IIIB) or metastatic (Stage IV) disease.
* Completion of 4 cycles of an acceptable, standard, platinum-based chemotherapy doublet without progression.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients of reproductive potential must agree to use effective contraception.

Exclusion Criteria:

* Prior exposure to agents directed at the human epidermal growth factor receptor (HER) axis (eg, gefitinib, cetuximab, trastuzumab).
* Prior treatment with any monoclonal antibody therapy.
* Any other malignancies within the previous 5 years, except for adequately treated carcinoma in situ of the cervix or squamous cell skin cancer.
* Clinically significant cardiovascular, hepatic, renal, or metabolic disease or active infection
* Pre-existing interstitial lung disease.
* Human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- India (7):
  - Bangalore
  - Chennai
  - Delhi
  - Hyderabad
  - Jaipur
  - Kolkata
  - Nashik

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib
Started | 51
Completed | 2
Not Completed | 49
Not completed — Disease Progression | 41
Not completed — Lost to Follow-up | 3
Not completed — Death | 4
Not completed — Withdrawal of Consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival at Week 52
Description: A participant had progression-free survival if they did not have disease progression and were alive. Tumor assessments were done by magnetic resonance imaging according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-target lesions. All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: From the date of enrolment in the study until the date of disease progression or death from any cause (up to 2 years, 6 months).
Population: Full analysis set: All enrolled participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 51
Percentage of participants | 22.5

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of enrolment to the date of disease progression (PD) or death, whichever occurred first. Tumor assessments were done by magnetic resonance imaging according to RECIST v1.1. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions (TL), taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-TLs. All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as TLs at Baseline. TLs should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all TLs will be calculated and reported as the Baseline sum longest diameter.
Time Frame: From the date of enrolment until the end of the study (up to 2 years, 6 months).
Population: Full analysis set: All enrolled participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Erlotinib
Number analyzed (Participants) | 51
Days | 99 [53.0 to 292.0]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of enrolment to the date of death from any cause.
Time Frame: From the date of enrolment until the end of the study (up to 2 years, 6 months).
Population: Full analysis set: All enrolled participants.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Erlotinib
Number analyzed (Participants) | 51
Days | 671 [392 to 796]

4. Secondary Outcome: Percentage of Participants With a Complete Response (CR) or a Partial Response (PR)
Description: A CR was defined as the disappearance of all target lesions. A PR was defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the Baseline sum longest diameter. All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. All other lesions (or sites of disease) should be identified as non-target lesions. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter. Tumor assessments were done by magnetic resonance imaging according to RECIST v1.1.
Time Frame: From the date of enrolment until the end of the study (up to 2 years, 6 months).
Population: Full analysis set: All enrolled participants. The analysis only included 47 participants as data for 4 participants was not available.
Measure: Number; unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 47
Percentage of participants
  Complete response | 2.1
  Partial response | 23.4

5. Secondary Outcome: Percentage of Participants With Disease Control
Description: A participant with disease control was defined as a participant with either a complete response (CR), a partial response (PR), or stable disease (SD), as determined using RECIST v1.1. A CR was defined as the disappearance of all target lesions (TL). A PR was defined as at least a 30% decrease in the sum of the longest diameter of TLs taking as reference the Baseline sum longest diameter (SLD). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest SLD since treatment started. For non-TLs, SD was defined as the persistence of 1 or more lesions. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since treatment started or the unequivocal progression of existing non-TLs. A SLD for all TLs will be calculated and reported as the Baseline SLD. Tumor assessments were done by magnetic resonance imaging according to RECIST v1.1.
Time Frame: From the date of enrolment until the end of the study (up to 2 years, 6 months).
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 47
Percentage of participants | 55.3

ADVERSE EVENTS:
Description: Safety population: All participants who had received at least 1 dose of erlotinib and had at least 1 safety follow-up, whether withdrawn prematurely or not.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 4/51
Other Adverse Events (participants affected / at risk) | 32/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=51)
Deep vein thrombosis (Vascular disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Convulsions (Nervous system disorders) | 1
Gastrointestinal toxicity (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=51)
Acneiform rash (Skin and subcutaneous tissue disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dyspnoea (Cardiac disorders) | 4
Fever (General disorders) | 3
Generalized weakness (General disorders) | 4
Headache (Nervous system disorders) | 3
Itching (Skin and subcutaneous tissue disorders) | 3
Maculopapular rashes (Skin and subcutaneous tissue disorders) | 3
Rashes (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.